CLINICAL TRIAL: NCT01105507
Title: An Open Label Study to Assess the Safety, Tolerability and Efficacy of Canakinumab (ACZ885) in Patients Aged 4 Years or Older Diagnosed With Cryopyrin-associated Periodic Syndromes (CAPS) in Canada
Brief Title: The Safety and Efficacy of Canakinumab in Patients Aged 4 Years or Older Diagnosed With Cryopyrin-associated Periodic Syndromes (CAPS) in Canada
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885DCA01
Record Dates: First submitted 2010-03-25; First posted 2010-04-16 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Cryopyrin Associated Periodic Syndrome
Keywords: Canakinumab; Cryopyrin-associated periodic syndromes; Familial Cold Autoinflammatory Syndrome (FCAS); Familial Cold Urticaria (FCU); Muckle-Wells Syndrome (MWS); Neonatal-Onset Multisystem Inflammatory Disease (NOMID); Chronic Infantile Neurological; Cutaneous; Articular Syndrome (CINCA); Treatment of patients diagnosed with CAPS (Cryopyrin associated periodic syndrome)
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — canakinumab

ARMS (1):
- canakinumab arm (Experimental)
  Interventions: Drug: canakinumab (company code: ACZ885D)

INTERVENTIONS:
Drug: canakinumab (company code: ACZ885D)

SUMMARY:
This study will assess the safety, tolerability and efficacy of canakinumab treatment in Canadian patient diagnosed with cryopyrin-associated periodic syndrome over a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients at least 4 years of age at the time of the screening visit
2. Patient's informed consent for > or = 18 years of age before any assessment is performed
3. Parent or legal guardian's written informed consent and child's assent, if appropriate, are required before any assessment is performed for patients < 18 years of age.
4. Patients with a diagnosis of CAPS: FCAS/FCU, MWS, or NOMID/CINCA
5. Body weight > or = 15 kg
6. Able to communicate with the investigator and comply with the requirements of the study (for children the parent can assist when necessary)

Exclusion Criteria:

1. Patient is pregnant or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test at baseline
2. Patient of childbearing potential (man or woman) and unwilling to use double barrier method of contraception. It is required that double barrier method of contraception be used (i.e. condom with spermicide or diaphragm with spermicide) by patients of childbearing potential (man or woman) regardless of whether a hormonal agent is also used as a method of contraception.
3. Participation in any clinical investigation within 4 weeks prior to dosing
4. Live vaccinations within 3 months prior to the start of the trial, during the trial and up to 3 months following the last dose.
5. History of significant medical conditions, which in the Investigator's opinion would exclude the patient from participating in this trial (this can be discussed with Novartis on a case by case basis in case of uncertainty).
6. History of drug or alcohol abuse within 12 months prior to dosing
7. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes

"Other protocol-defined inclusion/exclusion criteria may apply"

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05-12 (Actual); Study Completion 2012-05-12 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability of canakinumab by measuring the maintenance of response over time using the Investigators Clinical Assessment of Disease Activity scale and the evaluation of serum inflammation markers CRP (C-Reactive Protein), SAA (Serum Amyloid A. | 18 months

SECONDARY OUTCOMES:
Change in long term maintenance of Health-Related Quality of Life and productivity measured from baseline to end of study. | Baseline, 18 months
Treatment adherence with canakinumab for the duration of the study. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Department of Pediatrics, Calgary
  - Queen Elizabeth II Hospital, Halifax